CLINICAL TRIAL: NCT01149655
Title: A Long-Term Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Aripiprazole (OPC 14597) as Maintenance Treatment in Adolescent Patients With Schizophrenia
Brief Title: Efficacy & Safety Study of Oral Aripiprazole in Adolescents With Schizophrenia
Acronym: ATTAIN 266
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 31-09-266
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: Adolescent; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1 (Experimental): Aripiprazole (2-mg, 5-mg, 10-mg, 15-mg, 20-mg, 25-mg or 30-mg)
  Interventions: Drug: Aripiprazole
- Phase 2 (Experimental): Aripiprazole (2-mg, 5-mg, 10-mg, 15-mg, 20-mg, 25-mg or 30-mg)
  Interventions: Drug: Aripiprazole
- Phase 3 (Placebo Comparator): Aripiprazole (10-mg, 15-mg, 20-mg, 25-mg or 30-mg) or placebo
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole (2-mg, 5-mg, 10-mg, 15-mg, 20-mg, 25-mg or 30-mg)
  Arms: Phase 1; Phase 2
Drug: Aripiprazole — Aripiprazole (10-mg, 15-mg, 20-mg, 25-mg or 30-mg)
  Arms: Phase 3

SUMMARY:
This will be a randomized, double-blind, placebo-controlled study consisting of a screening period, a conversion phase (Phase 1), a stabilization phase (Phase 2), and a double-blind maintenance treatment phase (Phase 3), and a follow up period.

Subjects may be either outpatients or inpatients between screening and through the time they reach stabilization at the end of Phase 2; hospitalization is not a study requirement. However, eligible subjects must be outpatients at the beginning of Phase 3.

Subjects will be assessed weekly during Phase 1, weekly for the first 4 weeks of Phase 2 and 3, and biweekly for the remaining weeks during each of Phases 2 and 3. Subjects will be encouraged to call the investigators with any exacerbation of psychotic symptoms and/or any tolerability issues. The investigator will also have the option to phone the subjects and their guardian(s) at any time to ensure clinical stability.

A data monitoring committee (DMC) will provide oversight for safety monitoring and reviewing the interim analysis. One interim analysis is planned after 75% of the total expected number of impending relapse events (28 events) are achieved and will be conducted by an independent data analysis center. The DMC will make a recommendation about stopping or continuing the study based on safety and efficacy reviews. The results of the interim analysis and individual subject data will remain blinded to the sponsor during the course of the study until the DMC determines that the study will conclude based on the results of the interim analysis, or the study is completed after 37 endpoint events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a current DSM-IV-TR diagnosis of schizophrenia, and a history of the illness (diagnosis or symptoms) for at least 6 months prior to screening.
* Subjects who have shown previous response to antipsychotic treatment (other than clozapine) and are not resistant to treatment with other antipsychotics.
* Subjects who are currently being treated with oral or depot antipsychotics other than clozapine.
* Subjects with a history of relapse and/or exacerbation of symptoms when they are not receiving antipsychotic treatment.

Exclusion Criteria:

* Subjects with a current DSM-IV-TR diagnosis other than schizophrenia.
* Subjects with delirium, dementia, amnesia or other cognitive disorders; subjects with psychotic symptoms that are better accounted for by another general medical condition(s) or direct effect of a substance (i.e., medication, illicit drug use, etc.).
* Subjects with attention deficit disorder or attention deficit hyperactivity disorder and/or subjects who were on a stimulant treatment for any period of time over the last one year prior to screening.
* Subjects with any neurodevelopmental disorder, except Tourette's syndrome.
* Subjects experiencing acute depressive symptoms within the past 30 days prior to screening.
* Subjects who meet the DSM-IV-TR criteria for substance dependence (including alcohol and benzodiazepines, but excluding caffeine and nicotine) within the past 180 days prior to screening.
* Subjects who have epilepsy, a history of seizures (except for a single childhood febrile seizure or post-traumatic seizure), or a history of severe head trauma or stroke, or have a history or current evidence of other unstable medical conditions.
* Subjects with a history of subclinical hypothyroidism (TSH ≥ 4.0 mIU/L), known hypothyroidism or hyperthyroidism (unless the condition has been stabilized with medication for at least 90 days prior to entry into Phase 1 or Phase 2).
* Subjects who have a medical history of uncontrolled diabetes, labile or unstable diabetes (brittle diabetes), newly diagnosed diabetes, or clinically significant abnormal blood glucose levels.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development and Commercialization, Inc.
Locations (50):
- United States (8):
  - Study Site, Downy, California
  - Study Site, Glendale, California
  - Study Site, Miami, Florida
  - Study Site, Miami Springs, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Bloomfield Hills, Michigan
  - Study Site, Chapel Hill, North Carolina
  - Study Site, Bothell, Washington
- India (11):
  - Study Site, Vijayawada, Andhra Pradesh
  - Study Site, Visakhapatnam, Andhra Pradesh
  - Study Site, Raipur, Chhattisgarh
  - Study Site, Maninagar, Ahmedabad, Gujarat
  - Study Site, Aurangabad, Maharashtra
  - Study Site, Wardha, Maharashtra
  - Study Site, Chennai, Tamil Nadu
  - Study Site, Madurai, Tamil Nadu
  - Study Site, Lucknow, Uttar Pradesh
  - Study Site, Varanasi, Uttar Pradesh
  - Study Site, Guntur
- Malaysia (4):
  - Study Site, Kuala Lumpur, Kuala Lumpur
  - Study Site, Ipoh, Perak
  - Study Site, Batu Caves, Selangor
  - Study Site, Johor Bahru
- Philippines (5):
  - Study Site, Dasmariñas, Cavite
  - Study Site, Bajada, Davao City
  - Study Site, Manila, National Capital Region
  - Study Site, Iloilo City
  - Study Site, Mandaluyong
- Romania (5):
  - Study Site, Cluj-Napoca, Cluj
  - Study Site, Craiova, Dolj
  - Study Site, Timișoara, Timiș County
  - Study Site, Bucharest
  - Study Site, Iași
- Russia (14):
  - Study Site, Arkhangelsk
  - Study Site, Kazan'
  - Study Site, Lipetsk
  - Study Site, Moscow
  - Study Site, Nizhny Novgorod
  - Study Site, Novosibirsk
  - Study Site, Orenburg
  - Study Site, Petrozavodsk
  - Study Site, Saint Petersburg
  - Study Site, Saratov
  - Study Site, Tomsk
  - Study Site, Tonnelnyi Township
  - Study Site, Yaroslavl
  - Study Site, Yekaterinburg
- Taiwan (3):
  - Study Site, Kaohsiung County
  - Study Site, Taipei
  - Study Site, Taoyuan

REFERENCES:
- [Derived] Correll CU, Kohegyi E, Zhao C, Baker RA, McQuade R, Salzman PM, Sanchez R, Nyilas M, Carson W. Oral Aripiprazole as Maintenance Treatment in Adolescent Schizophrenia: Results From a 52-Week, Randomized, Placebo-Controlled Withdrawal Study. J Am Acad Child Adolesc Psychiatry. 2017 Sep;56(9):784-792. doi: 10.1016/j.jaac.2017.06.013. Epub 2017 Jul 8. PMID 28838583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase 3 randomized, double-blind, placebo-controlled study consisted of screening period, conversion (Period 1), stabilization (Period 2), double-blind maintenance treatment (Period 3) and a follow-up period to evaluate efficacy and safety of aripiprazole (10-30 mg/day) compared to placebo in adolescent participants with schizophrenia.
Pre-assignment Details: Participants were titrated to oral aripiprazole in Period 1. Participants who converted to aripiprazole and who already received aripiprazole were in Period 2. Participants met stability criteria were randomized in 2:1 ratio (aripiprazole: placebo) in Period 3. 244 participants were screened of which 201 entered the trial and 146 were randomized.
Groups:
- Aripiprazole-Conversion Phase: Participants who had received oral aripiprazole 2 to 10 mg for 2 Weeks in combination with any other antipsychotic were in conversion phase.
- Aripiprazole-Stabilization Phase: Participants who had converted to aripiprazole monotherapy period 1 (conversion phase) and had received aripiprazole monotherapy for schizophrenia at screening were in period 2, provided the prescribed aripiprazole dose did not exceed 30 mg (milligrams) per day for 2 Weeks.
- Aripiprazole-Double Blind (DB) Maintenance: Participants who met stability criteria in period 2 (stabilization phase) received oral aripiprazole 10 to 30 mg/day for 52 Weeks in period 3 (double-blind maintenance treatment).
- Aripiprazole-Placebo-DB Maintenance: Participants who met stability criteria in period 2 (stabilization phase) received placebo for 52 Weeks in period 3 (double-blind maintenance treatment).
Period: Period 1 - Conversion Phase
Arm/Group | Aripiprazole-Conversion Phase | Aripiprazole-Stabilization Phase | Aripiprazole-Double Blind (DB) Maintenance | Aripiprazole-Placebo-DB Maintenance
Started | 186 | 0 | 0 | 0
Completed | 168 | 0 | 0 | 0
Not Completed | 18 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Sponsor Discontinued Trial | 4 | 0 | 0 | 0
Not completed — Met Withdrawal Criteria | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 0
Not completed — Adverse Event Without Relapse | 3 | 0 | 0 | 0
Period: Period 2-Stabilization Phase
Arm/Group | Aripiprazole-Conversion Phase | Aripiprazole-Stabilization Phase | Aripiprazole-Double Blind (DB) Maintenance | Aripiprazole-Placebo-DB Maintenance
Started | 0 | 183 | 0 | 0
Completed | 0 | 146 | 0 | 0
Not Completed | 0 | 37 | 0 | 0
Not completed — Sponsor Discontinued Trial | 0 | 16 | 0 | 0
Not completed — Met Withdrawal Criteria | 0 | 7 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 0 | 0
Not completed — Adverse Event Without Relapse | 0 | 6 | 0 | 0
Period: Period 3-DB Maintenance Phase
Arm/Group | Aripiprazole-Conversion Phase | Aripiprazole-Stabilization Phase | Aripiprazole-Double Blind (DB) Maintenance | Aripiprazole-Placebo-DB Maintenance
Started | 0 | 0 | 98 | 48
Completed | 0 | 0 | 15 | 6
Not Completed | 0 | 0 | 83 | 42
Not completed — Sponsor Discontinued Trial | 0 | 0 | 58 | 19
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 4
Not completed — Adverse Event Without Relapse | 0 | 0 | 1 | 1
Not completed — Relapse With AE | 0 | 0 | 19 | 18

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole-Double Blind Maintenance: Participants in period 3 were randomized in a 2:1 (aripiprazole: placebo) ratio and had received oral aripiprazole in the range of 10 to 30 mg/day as double-blind maintenance treatment for up to 52 weeks.
- Placebo-Double Blind Maintenance: Participants in period 3 were randomized in a 2:1 (aripiprazole: placebo) ratio and had received placebo as double-blind maintenance treatment for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance | Total
Number analyzed (Participants) | 98 | 48 | 146
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Male | 15.3 (1.3) | 15.6 (1.1) | 15.4 (1.2)
  Female | 15.4 (1.1) | 15.3 (1.0) | 15.3 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 14 | 50
  Male | 62 | 34 | 96

OUTCOME MEASURES:

1. Primary Outcome: Overall Relapse Rate (in Percent) From Randomization to Exacerbation of Psychotic Symptoms/Impending Relapse.
Description: The primary efficacy variable was overall relapse rate from randomization, as assessed by Clinical Global Impression of Improvement (CGI-I) score ≥5, Positive and Negative Syndrome Scale (PANSS) scores for hostility or uncooperativeness ≥5, or ≥20% increase in PANSS Total Score. Impending relapse was defined as meeting any of the following 5 criteria: 1) CGI-I score of ≥ 5 (minimally worse) and increase in individual PANSS items to a score > 4 with an absolute increase of ≥ 2 on that specific item or absolute increase of ≥ 4 on the combined 4 PANSS items (conceptual disorganization, hallucinatory behavior, suspiciousness, unusual thought content). OR 2) CGI-I score of 6 or 7 (much or very much worse) OR 3) Hospitalization due to worsening of illness OR 4) Any suicidal behavior or answers of "yes" to Questions 4 or 5 on the suicidal ideation section of the C-SSRS OR 5) Violent or aggressive behavior resulting in clinically significant injury.
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: For the primary analysis, participants that belonged to the ITT (intent to treat) data set were included in the analysis. Participants who were lost to follow-up or who were still in the study at the end of Week 52 were considered as censored on their date of last efficacy evaluation. The ITT data set comprised participants randomized to period 3.
Measure: Number; unit: relapse rate(percentage of participants)
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
relapse rate(percentage of participants) | 19.39 | 37.50
Statistical Analysis 1: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; The total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0161, Log Rank; The log-rank test was based on time to exacerbation of psychotic symptoms/impending relapse; Cox Proportional Hazard = 0.461, 95% CI 2-sided [0.242 to 0.879] — Hazard ratios and their 95% confidence intervals were derived from the Cox Proportional Hazard model with treatment as term. Hazard ratio < 1 is in favor of oral aripiprazole 10-30 mg group for superiority test

2. Secondary Outcome: Percentage of Participants Meeting Exacerbation of Psychotic Symptoms/Impending Relapse Criteria.
Description: Impending relapse was defined as meeting any of the following 5 criteria: 1) CGI-I score of ≥ 5 (minimally worse) and increase in individual PANSS items to a score > 4 with an absolute increase of ≥ 2 on that specific item or absolute increase of ≥ 4 on the combined 4 PANSS items. OR 2) CGI-I score of 6 or 7 (much or very much worse) OR 3) Hospitalization due to worsening of illness OR 4) Any suicidal behavior or answers of "yes" to Questions 4 or 5 on the suicidal ideation section of the C-SSRS OR 5) Violent or aggressive behavior resulting in clinically significant injury.
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: The ITT data set comprised of all participants who were randomized to period 3.
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
percentage of participants
  CGI-I + PANSS | 16.33 | 33.33
  CGI-I of 6 or 7 | 11.22 | 25.00
  Hospitalization | 1.02 | 10.42
  Suicidal Behavior | 1.02 | 0.00
  Violent Behavior | 4.08 | 10.42

3. Secondary Outcome: Percentage of Responders in Each Treatment Group.
Description: Percentage of responders in each treatment group (i.e, response defined as meeting stability criteria). Participants stabilized on aripiprazole (trial drug) within the approved dose range of 10 to 30 mg/day and are tolerable based on clinical judgment.
Time Frame: Baseline to Week 52/End of Phase 3 visit
Population: The ITT data set comprised of all participants were randomized to period 3.
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
percentage of participants
  Week 1 (Arirpiprazole N= 95, Placebo N= 45) | 96.8 | 97.8
  Week 2 (N= 91, 46) | 92.3 | 95.7
  Week 3 (N= 86, 45) | 93.0 | 86.7
  Week 4 (N= 91, 43) | 93.4 | 90.7
  Week 6 (N= 87, 41) | 90.8 | 92.7
  Week 8 (N= 82, 38) | 97.6 | 89.5
  Week 10 (N= 74, 32) | 94.6 | 93.8
  Week 12 (N= 71, 30) | 94.4 | 93.3
  Week 14 (N= 68, 26) | 94.1 | 92.3
  Week 16 (N= 65, 25) | 96.9 | 96.0
  Week 18 (N= 59, 23) | 94.9 | 91.3
  Week 20 (N= 57, 23) | 94.7 | 91.3
  Week 22 (N= 55, 21) | 92.7 | 95.2
  Week 24 (N= 51, 19) | 98.0 | 100.0
  Week 26 (N= 48, 19) | 97.9 | 100.0
  Week 28 (N= 42, 17) | 97.6 | 100.0
  Week 30 (N= 40, 16) | 95.0 | 100.0
  Week 32 (N= 39, 16) | 94.9 | 93.8
  Week 34 (N= 38, 14) | 94.7 | 100.0
  Week 36 (N= 36, 15) | 94.4 | 100.0
  Week 38 (N= 33, 12) | 100.0 | 100.0
  Week 40 (N= 29, 11) | 100.0 | 100.0
  Week 42 (N= 27, 11) | 100.0 | 100.0
  Week 44 (N= 21, 8) | 100.0 | 100.0
  Week 46 (N= 18, 8) | 88.9 | 100.0
  Week 48 (N= 17, 8) | 94.1 | 100.0
  Week 50 (N= 17, 6) | 88.2 | 100.0
  Week 52 (N= 14, 7) | 100.0 | 100.0
  Last Visit (N= 98, 48) | 77.6 | 64.6
Statistical Analysis 1: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical Analysis for Last Visit. The total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0962, Chi-squared; p-value was derived using Chi-square test

4. Secondary Outcome: Percentage of Participants Who Had Achieved Remission.
Description: Percentage of participants who had achieved remission, where remission was defined as a score of ≤ 3 on each of the following specific PANSS items, maintained for a period of 6 months: delusions, unusual thought content, hallucinatory behavior, conceptual disorganization, mannerisms/ posturing, blunted affect, social withdrawal, and lack of spontaneity.
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: The ITT data set comprised of participants who were randomized to the double-blind treatment. For evaluation of remission, 48 of 98 aripiprazole participants and 19 of 48 placebo participants met the 6 month threshold for remission analysis. Of those, 21 of 48 aripiprazole participants and 8 of 19 placebo participants met criteria for remission.
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 48 | 19
percentage of participants | 43.8 | 42.1
Statistical Analysis 1: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.9025, Chi-squared; p-value was derived using Chi-square test

5. Secondary Outcome: Percentage of Participants Who Discontinued Due to All Reasons Other Than Sponsor Discontinued Study.
Description: Percentage of participants discontinued due to all reasons other than sponsor discontinued study were noted.
Time Frame: Baseline to Week 52/End of Phase 3 visit
Population: The ITT data set comprised of all participants who were randomized to period 3.
Measure: Number; unit: percentage of participants
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
percentage of participants | 25.51 | 47.92
Statistical Analysis 1: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0076, Log Rank; p-value was derived from the log-rank tests

6. Other Pre Specified Outcome: Mean Change From Baseline to Endpoint in PANSS Total Score.
Description: The PANSS consisted of 3 subscales with a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicates (absence of symptoms) and a score of 7 indicates (extremely severe symptoms). The symptom constructs for each subscale were positive subscale, negative subscale and general psychopathology subscale. The PANSS Total Score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: The ITT data set comprised of participants randomized to period 3. LOCF (last observation carried forward) method was used to impute missing data. Week 1 had only 95 and 45 participants analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
Units on a scale
  Week 1 (Aripiprazole N= 95, Placebo N= 45) | 0.22 (5.62) | -0.27 (4.66)
  Week 2 | 0.09 (5.77) | -0.58 (6.01)
  Week 3 | -0.36 (6.41) | 1.81 (9.66)
  Week 4 | -0.64 (6.90) | 1.56 (11.13)
  Week 6 | -1.20 (8.28) | 2.92 (13.39)
  Week 8 | -1.62 (9.20) | 3.71 (14.29)
  Week 10 | -1.20 (9.61) | 3.90 (14.80)
  Week 12 | -0.19 (10.57) | 4.52 (16.17)
  Week 14 | -0.18 (11.06) | 5.50 (17.21)
  Week 16 | -0.78 (11.72) | 5.56 (17.33)
  Week 18 | -0.68 (12.30) | 5.57 (17.24)
  Week 20 | -0.57 (12.46) | 6.06 (17.84)
  Week 22 | -0.31 (12.37) | 6.10 (18.98)
  Week 24 | -0.36 (12.36) | 5.92 (19.22)
  Week 26 | -0.88 (12.41) | 5.81 (19.65)
  Week 28 | -0.85 (12.52) | 5.65 (19.82)
  Week 30 | -0.96 (12.71) | 5.60 (19.96)
  Week 32 | -0.99 (12.74) | 6.21 (20.43)
  Week 34 | -1.12 (13.05) | 5.79 (19.85)
  Week 36 | -0.55 (13.04) | 5.40 (20.20)
  Week 38 | -0.84 (13.17) | 5.21 (20.27)
  Week 40 | -0.92 (13.21) | 5.10 (20.34)
  Week 42 | -1.14 (13.26) | 4.94 (20.36)
  Week 44 | -0.96 (13.32) | 4.88 (20.47)
  Week 46 | -1.02 (13.35) | 4.83 (20.54)
  Week 48 | -0.99 (13.34) | 4.67 (20.72)
  Week 50 | -1.19 (13.43) | 4.71 (20.66)
  Week 52 | -1.31 (13.47) | 4.79 (20.60)

7. Other Pre Specified Outcome: Mean Change From Baseline to Endpoint in CGI-S Score.
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-s, the Investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0= not assessed; 1= normal, not at all ill; 2= borderline mentally ill; 3= mildly ill; 4= moderately ill; 5= markedly ill; 6= severely ill; and 7= among the most extremely ill participants.
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: The ITT data set comprised of participants randomized to period 3. LOCF method was used to impute missing data. Week 1 participants analyzed were 94 and 45 and Week 2 to Week 52 participants analyzed were 97 and 48.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
Units on a scale
  Week 1 (Aripiprazole N= 94, Placebo N= 45) | 0.01 (0.23) | 0.02 (0.34)
  Week 2 (N= 97, 48) | 0.00 (0.32) | 0.02 (0.44)
  Week 3 | 0.01 (0.40) | 0.13 (0.64)
  Week 4 | 0.03 (0.44) | 0.10 (0.69)
  Week 6 | 0.04 (0.52) | 0.15 (0.77)
  Week 8 | 0.04 (0.63) | 0.19 (0.79)
  Week 10 | 0.02 (0.71) | 0.25 (0.81)
  Week 12 | 0.05 (0.77) | 0.31 (0.85)
  Week 14 | 0.03 (0.78) | 0.35 (1.04)
  Week 16 | 0.02 (0.83) | 0.33 (1.06)
  Week 18 | 0.04 (0.83) | 0.35 (1.06)
  Week 20 | 0.05 (0.85) | 0.40 (1.12)
  Week 22 | 0.08 (0.87) | 0.38 (1.14)
  Week 24 | 0.06 (0.88) | 0.35 (1.18)
  Week 26 | 0.05 (0.89) | 0.35 (1.18)
  Week 28 | 0.05 (0.92) | 0.33 (1.19)
  Week 30 | 0.04 (0.91) | 0.33 (1.19)
  Week 32 | 0.04 (0.92) | 0.31 (1.21)
  Week 34 | 0.05 (0.93) | 0.29 (1.22)
  Week 36 | 0.07 (0.95) | 0.29 (1.22)
  Week 38 | 0.07 (0.95) | 0.29 (1.22)
  Week 40 | 0.07 (0.95) | 0.29 (1.22)
  Week 42 | 0.06 (0.94) | 0.29 (1.22)
  Week 44 | 0.08 (0.95) | 0.31 (1.21)
  Week 46 | 0.07 (0.95) | 0.31 (1.21)
  Week 48 | 0.06 (0.94) | 0.29 (1.22)
  Week 50 | 0.05 (0.95) | 0.27 (1.25)
  Week 52 | 0.05 (0.95) | 0.29 (1.22)

8. Other Pre Specified Outcome: Mean CGI-I Score at Endpoint.
Description: Baseline for the double-blind maintenance phase was defined as the last visit with available data in the stabilization phase, and the CGI-I scale was completed prior to or on the first dose date in the double-blind maintenance phase. Response choices included: 0 = not assessed; 1 = very much improved,;2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
Units on a scale
  Baseline | 2.40 (0.80) | 2.52 (0.82)
  Week 1 (Aripiprazole N= 94, Placebo N= 45) | 3.49 (0.84) | 3.51 (0.84)
  Week 2 (N= 97, 48) | 3.48 (0.88) | 3.52 (0.95)
  Week 3 | 3.47 (0.89) | 3.63 (1.06)
  Week 4 | 3.60 (0.92) | 3.60 (1.20)
  Week 6 | 3.53 (1.00) | 3.73 (1.30)
  Week 8 | 3.46 (1.09) | 3.83 (1.45)
  Week 10 | 3.38 (1.13) | 3.90 (1.49)
  Week 12 | 3.45 (1.19) | 3.96 (1.44)
  Week 14 | 3.44 (1.23) | 4.04 (1.56)
  Week 16 | 3.32 (1.25) | 4.00 (1.57)
  Week 18 | 3.35 (1.29) | 4.02 (1.58)
  Week 20 | 3.40 (1.30) | 4.08 (1.54)
  Week 22 | 3.43 (1.34) | 4.04 (1.60)
  Week 24 | 3.41 (1.31) | 4.06 (1.60)
  Week 26 | 3.41 (1.34) | 4.06 (1.60)
  Week 28 | 3.43 (1.34) | 4.02 (1.64)
  Week 30 | 3.44 (1.36) | 4.00 (1.66)
  Week 32 | 3.46 (1.37) | 3.98 (1.68)
  Week 34 | 3.47 (1.36) | 3.94 (1.71)
  Week 36 | 3.48 (1.39) | 3.94 (1.71)
  Week 38 | 3.45 (1.38) | 3.94 (1.71)
  Week 40 | 3.45 (1.38) | 3.92 (1.72)
  Week 42 | 3.45 (1.38) | 3.92 (1.72)
  Week 44 | 3.45 (1.38) | 3.94 (1.71)
  Week 46 | 3.46 (1.37) | 3.94 (1.71)
  Week 48 | 3.46 (1.38) | 3.92 (1.72)
  Week 50 | 3.43 (1.38) | 3.92 (1.72)
  Week 52 | 3.42 (1.39) | 3.92 (1.72)
Statistical Analysis 1: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis at Baseline. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.3862, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 2: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 1. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.8861, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 3: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 2. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.8189, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 4: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 3. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.3689, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 5: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 4. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.9723, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 6: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 6. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.2985, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 7: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 8. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0883, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 8: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 10. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0228, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 9: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 12. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0274, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 10: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 14. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0135, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 11: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 16. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0059, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 12: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 18. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0076, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 13: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 20. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0065, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 14: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 22. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0175, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 15: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 24. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0107, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 16: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 26. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0118, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 17: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 28. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0232, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 18: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 30. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0337, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 19: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 32. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0507, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 20: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 34. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0791, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 21: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 36. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0898, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 22: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 38. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0686, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 23: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 40. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0833, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 24: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 42. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0824, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 25: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 44. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0686, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 26: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 46. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0737, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 27: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 48. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0893, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 28: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 50. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0706, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics
Statistical Analysis 29: Comparison: Aripiprazole-Double Blind Maintenance vs Placebo-Double Blind Maintenance; Statistical analysis for Week 52. The expected total number of exacerbation of psychotic symptoms/impending relapse was estimated using a 2:1 (aripiprazole:placebo) randomization ratio to achieve at least 80% power and to preserve an overall nominal alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0657, Cochran-Mantel-Haenszel; CMH method was based on raw mean score statistics

9. Other Pre Specified Outcome: Mean Change From Baseline to Endpoint in PANSS Positive Subscale.
Description: The PANSS consisted of 3 subscales were a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicated (absence of symptoms) and a score of 7 indicated (extremely severe symptoms). The 7 positive symptom constructs were delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS Total Score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: The ITT data set comprised of participants randomized to period 3. LOCF method was used to impute missing data. Week 1 participants analyzed were 94 and 45.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
Units on a scale
  Week 1 (Aripiprazole N= 95, Placebo N= 45) | 0.08 (1.84) | 0.07 (2.41)
  Week 2 | 0.09 (2.05) | -0.04 (2.87)
  Week 3 | 0.01 (2.36) | 0.56 (3.34)
  Week 4 | -0.12 (2.65) | 0.58 (3.80)
  Week 6 | -0.20 (2.90) | 1.10 (4.85)
  Week 8 | -0.19 (3.23) | 1.56 (5.11)
  Week 10 | -0.16 (3.28) | 1.63 (5.45)
  Week 12 | 0.23 (3.58) | 1.96 (5.78)
  Week 14 | 0.28 (3.77) | 2.27 (6.03)
  Week 16 | 0.32 (3.77) | 2.17 (6.05)
  Week 18 | 0.24 (3.98) | 2.15 (6.14)
  Week 20 | 0.18 (4.00) | 2.44 (6.32)
  Week 22 | 0.39 (4.12) | 2.60 (6.44)
  Week 24 | 0.38 (4.23) | 2.65 (6.36)
  Week 26 | 0.22 (4.23) | 2.58 (6.45)
  Week 28 | 0.17 (4.28) | 2.56 (6.51)
  Week 30 | 0.24 (4.43) | 2.60 (6.59)
  Week 32 | 0.22 (4.41) | 2.71 (6.64)
  Week 34 | 0.18 (4.45) | 2.58 (6.54)
  Week 36 | 0.29 (4.45) | 2.48 (6.60)
  Week 38 | 0.22 (4.55) | 2.46 (6.63)
  Week 40 | 0.27 (4.56) | 2.44 (6.69)
  Week 42 | 0.24 (4.52) | 2.35 (6.73)
  Week 44 | 0.27 (4.52) | 2.33 (6.76)
  Week 46 | 0.21 (4.52) | 2.42 (6.69)
  Week 48 | 0.30 (4.53) | 2.29 (6.77)
  Week 50 | 0.20 (4.52) | 2.33 (6.75)
  Week 52 | 0.16 (4.55) | 2.31 (6.77)

10. Other Pre Specified Outcome: Mean Change From Baseline to Endpoint in PANSS Negative Subscale.
Description: The PANSS consisted of 3 subscales were a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicated (absence of symptoms) and a score of 7 indicated (extremely severe symptoms). The 7 negative symptom constructs were blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation and stereotyped thinking. The PANSS Total Score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
Units on a scale
  Week 1 (Aripiprazole N= 95, Placebo N= 45) | 0.03 (1.57) | -0.09 (1.40)
  Week 2 | -0.07 (1.68) | -0.23 (2.35)
  Week 3 | -0.39 (1.89) | 0.48 (3.17)
  Week 4 | -0.27 (2.12) | 0.44 (3.41)
  Week 6 | -0.42 (2.37) | 0.90 (3.57)
  Week 8 | -0.41 (2.37) | 0.77 (3.76)
  Week 10 | -0.33 (2.47) | 0.71 (3.82)
  Week 12 | -0.38 (2.91) | 0.79 (4.47)
  Week 14 | -0.41 (3.13) | 1.15 (4.63)
  Week 16 | -0.51 (3.31) | 1.19 (4.77)
  Week 18 | -0.47 (3.45) | 1.19 (4.75)
  Week 20 | -0.47 (3.54) | 1.10 (4.93)
  Week 22 | -0.43 (3.55) | 1.06 (5.26)
  Week 24 | -0.42 (3.54) | 0.79 (5.41)
  Week 26 | -0.54 (3.60) | 0.81 (5.43)
  Week 28 | -0.51 (3.63) | 0.83 (5.43)
  Week 30 | -0.56 (3.57) | 0.67 (5.55)
  Week 32 | -0.52 (3.60) | 0.98 (5.89)
  Week 34 | -0.64 (3.68) | 0.56 (5.61)
  Week 36 | -0.47 (3.71) | 0.65 (5.69)
  Week 38 | -0.62 (3.70) | 0.54 (5.84)
  Week 40 | -0.64 (3.78) | 0.54 (5.78)
  Week 42 | -0.77 (3.79) | 0.42 (5.75)
  Week 44 | -0.72 (3.87) | 0.46 (5.76)
  Week 46 | -0.68 (3.84) | 0.35 (5.83)
  Week 48 | -0.73 (3.83) | 0.33 (5.88)
  Week 50 | -0.80 (3.84) | 0.29 (5.96)
  Week 52 | -0.78 (3.81) | 0.40 (5.87)

11. Other Pre Specified Outcome: Mean Change From Baseline to Endpoint in Children's Global Assessment Scale (CGAS).
Description: The CGAS was developed by Schaffer and colleagues to provide a global measure of severity of disturbance in children and adolescents. The CGAS is a rating scale for evaluating the overall functioning of a participant during a specified time period on a continuum from psychological or psychiatric sickness to health. The CGAS is a valid and reliable tool for rating a child's general level of functioning on a health-illness continuum. CGAS score (range 1-100) was a single item score for rating a child's general level of functioning on a health-illness continuum, with higher scores represented better functioning.
Time Frame: Baseline to Week 52/End of Phase 3 visit.
Population: The ITT data set comprised of participants randomized to period 3. LOCF method was used to impute missing data. Week 1 participants analyzed were 95 and 45.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole-Double Blind Maintenance | Placebo-Double Blind Maintenance
Number analyzed (Participants) | 98 | 48
Units on a scale
  Week 1 (Aripiprazole N= 95, Placebo N= 45) | 0.00 (2.74) | -0.09 (2.02)
  Week 2 | -0.10 (3.90) | -0.31 (4.03)
  Week 3 | 0.35 (4.36) | -1.04 (7.21)
  Week 4 | 0.29 (5.22) | -1.23 (7.78)
  Week 6 | 0.40 (6.01) | -2.08 (9.14)
  Week 8 | 0.98 (6.90) | -2.40 (9.93)
  Week 10 | 1.11 (7.47) | -2.31 (11.63)
  Week 12 | 1.08 (8.21) | -2.85 (11.40)
  Week 14 | 1.06 (8.49) | -3.52 (12.40)
  Week 16 | 1.57 (8.69) | -2.69 (12.96)
  Week 18 | 1.55 (9.41) | -2.90 (13.07)
  Week 20 | 1.28 (9.88) | -4.06 (14.84)
  Week 22 | 1.17 (10.15) | -3.77 (15.05)
  Week 24 | 1.33 (10.33) | -3.67 (15.20)
  Week 26 | 1.61 (10.37) | -3.69 (15.29)
  Week 28 | 1.73 (10.73) | -3.75 (15.26)
  Week 30 | 1.92 (10.89) | -3.44 (15.45)
  Week 32 | 1.86 (11.03) | -3.33 (15.47)
  Week 34 | 2.05 (11.19) | -3.00 (15.85)
  Week 36 | 1.87 (11.41) | -3.10 (15.70)
  Week 38 | 2.00 (11.59) | -2.85 (15.95)
  Week 40 | 1.90 (11.68) | -2.85 (15.99)
  Week 42 | 1.90 (11.74) | -2.69 (16.17)
  Week 44 | 1.83 (11.86) | -2.67 (16.18)
  Week 46 | 2.13 (11.74) | -2.67 (16.17)
  Week 48 | 2.17 (11.79) | -2.40 (16.42)
  Week 50 | 2.29 (11.74) | -2.31 (16.51)
  Week 52 | 2.35 (11.85) | -2.25 (16.58)

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time the ICF was signed (with 4-Week Post-Trial Follow-up).
Description: A SAE was any untoward medical occurrence that results in death or was life-threatening or required inpatient hospitalization or prolonged hospitalization. An AE was an exacerbation of an existing problem or any new problem, experienced by a participant when enrolled in a trial, whether or not it was considered drug related by the study physician.
Groups:
- Aripiprazole-Conversion Phase: Participants had received oral aripiprazole 2 to 10 mg for 2 Weeks in combination with any other antipsychotic were in conversion phase.
- Arpiprazole-Stabilization Phase: Participants who had converted to aripiprazole monotherapy period 1 (conversion phase) and had received aripiprazole monotherapy for schizophrenia at screening were in period 2, provided the prescribed aripiprazole dose did not exceed 30 mg (milligrams) per day for 2 Weeks.
- Aripiprazole-Double Blind Maintenance Treatment: Participants who met stability criteria in period 2 (stabilization phase) had received oral aripiprazole 10 to 30 mg/day for 52 Weeks in period 3 (double-blind maintenance treatment).
- Placebo-Double Blind Maintenance Treatment: Participants who met stability criteria in period 2 (stabilization phase) had received placebo for 52 Weeks in period 3 (double-blind maintenance treatment).
Arm/Group | Aripiprazole-Conversion Phase | Arpiprazole-Stabilization Phase | Aripiprazole-Double Blind Maintenance Treatment | Placebo-Double Blind Maintenance Treatment
Serious Adverse Events (participants affected / at risk) | 0/186 | 4/183 | 3/98 | 6/48
Other Adverse Events (participants affected / at risk) | 52/186 | 56/183 | 41/98 | 25/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole-Conversion Phase (N=186) | Arpiprazole-Stabilization Phase (N=183) | Aripiprazole-Double Blind Maintenance Treatment (N=98) | Placebo-Double Blind Maintenance Treatment (N=48)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 2 | 1
Schizophrenia (Psychiatric disorders) | 0 | 2 | 1 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole-Conversion Phase (N=186) | Arpiprazole-Stabilization Phase (N=183) | Aripiprazole-Double Blind Maintenance Treatment (N=98) | Placebo-Double Blind Maintenance Treatment (N=48)
Akathisia (Nervous system disorders) | 11 | 14 | 3 | 3
Headache (Nervous system disorders) | 12 | 13 | 6 | 4
Insomnia (Psychiatric disorders) | 16 | 14 | 5 | 9
Nasopharyngitis (Infections and infestations) | 0 | 0 | 7 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 7 | 4
Schizophrenia (Psychiatric disorders) | 0 | 0 | 9 | 8
Somnolence (Nervous system disorders) | 19 | 12 | 0 | 0
Tremor (Nervous system disorders) | 0 | 13 | 4 | 4
Weight increased (Investigations) | 0 | 13 | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No